CLINICAL TRIAL: NCT04737330
Title: A Two-year Multi-center Phase 3 Study to Investigate the Efficacy and Safety of Secukinumab in Adult Patients With Active, Moderate to Severe Thyroid Eye Disease (ORBIT), With a Randomized, Parallel-group, Double-blind, Placebo-controlled, 16-week Treatment Period, and a Follow-up/Retreatment Period
Brief Title: A Study of the Efficacy and Safety of Secukinumab 300 mg in Patients With Thyroid Eye Disease (TED)
Acronym: ORBIT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Analysis of blinded patient data showed a very low probability of the study meeting the primary efficacy endpoints. No safety concerns were identified
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457ADE16; 2020-001611-24 (EudraCT Number)
Record Dates: First submitted 2020-11-20; First posted 2021-02-03 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Eye Disease; Graves Orbitopathy
Keywords: TED; Bulging eyes; Exophthalmos
MeSH Terms: conditions — Graves Ophthalmopathy; Exophthalmos | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secukinumab 300 mg (Active Comparator): Secukinumab 300 mg subcutaneous (s.c.) injection at Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12
  Interventions: Drug: Secukinumab
- Placebo (Placebo Comparator): Placebo subcutaneous (s.c.) injection at Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab — Secukinumab 300 mg s.c. at Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12
  Other Names: AIN457
  Arms: Secukinumab 300 mg
Drug: Placebo — Placebo s.c. at Baseline, Weeks 1, Week 2, Week 3, Week 4, Week 8, Week 12
  Arms: Placebo

SUMMARY:
Thyroid eye disease (TED) is a rare autoimmune, inflammatory disorder of the orbit and represents the most common extra-thyroidal manifestation of Graves' disease (GD). Several lines of evidence suggest an important role of interleukin-17A (IL-17A) in the pathogenesis of TED; increased levels of IL-17A have been detected in the serum and tears of patients with TED and IL-17A levels correlate with clinical activity of the disease. T-helper 17 cells (Th17 cells) (as well as other cellular sources of IL-17A, e.g., Tc17 cells) have been shown to infiltrate the orbital tissue of affected patients, producing IL-17A. IL-17A stimulates fibroblast activation, leading to retrobulbar tissue expansion and orbital fibrosis, which causes significant functional impairment. Secukinumab is a recombinant high-affinity fully human monoclonal anti-IL-17A antibody currently approved for the treatment of 3 inflammatory/ autoimmune diseases: moderate to severe plaque psoriasis (PsO), psoriatic arthritis (PsA), and axial spondyloarthritis (axSpA) (ankylosing spondylitis (AS) and non-radiographic axSpA). The purpose of this study was to demonstrate the efficacy and safety of secukinumab 300 mg subcutaneous (s.c.) in adults with active, moderate to severe TED.

DETAILED DESCRIPTION:
This study consisted of the following 3 periods:

1. Screening period (Week -6 to Baseline):

   Participants' eligibility was assessed during the Screening period, which occurred for a maximum of 6 weeks.
2. Treatment period (Baseline to Week 16):

   Eligible participants were randomized in a 1:1 ratio to one of the following double-blinded treatment arms:
   * Arm 1: Secukinumab 300 mg s.c. at Baseline, Week 1, 2, 3, 4, 8, 12
   * Arm 2: Placebo s.c. at Baseline, Week 1, 2, 3, 4, 8, 12

   Participants were stratified according to current smoking status (up to 20% smokers per arm) since smoking has a well-known impact on treatment efficacy in TED.
3. Follow-up/open-label retreatment period (Week 16 up to Week 108):

   * Proptosis responders (see definition below) at Week 16 were followed for relapse up to Week 68. If these participants relapsed, they were offered a course of open-label secukinumab at the time of relapse (see "proptosis relapsers" definition below).
   * Proptosis non-responders (see definition below) at Week 16 were offered the option of open-label secukinumab treatment (with maintenance of blind to initial randomized treatment) for a duration of 16 weeks, i.e., up to Week 32 with last dose at Week 28, as follows:

     * Open-label secukinumab 300 mg s.c. at Week 16, 17, 18, 19, 20, 24 and 28. Thereafter (i.e., from Week 32), participants were followed up for a further 24 weeks to assess the relapse rate.
     * For participants who were proptosis non-responders and who did not receive open-label secukinumab treatment, a follow-up visit 8 weeks after the Week 16 visit needed to be scheduled per protocol. At this follow-up visit, the assessments associated with the Week 24 visit (for responders) were to be performed.
   * Proptosis relapsers (see definition below) during the follow-up period (from Week 16 onward to Week 68) were offered the option of retreatment with open-label secukinumab for a duration of 16 weeks (with maintenance of blind to initial randomized treatment) at the time of relapse as follows:

     * Open-label secukinumab 300 mg s.c. at time of relapse, then at 1, 2, 3, 4, 8 and 12 weeks since time of relapse. Thereafter, participants were followed up for a further 24 weeks (i.e., 40 weeks after start of retreatment) to assess rate of relapse and safety.
     * For participants not receiving open-label secukinumab treatment a follow-up visit 8 weeks after the Week 16 visit were to be scheduled per protocol, if not yet completed. At this follow-up visit, the assessments associated with the Week 24 visit (for responders) were to be performed.

Definitions of proptosis responder, non-responder and relapser:

* Proptosis responders: Participants achieving response in reduction of proptosis at Week 16 defined as follows: reduction of >= 2 mm from Baseline in the study eye without deterioration (>= 2 mm increase) of proptosis in the fellow eye.
* Proptosis non-responders: Participants not achieving response in reduction of proptosis at Week 16 with "response" defined as follows: reduction of >= 2 mm from Baseline in the study eye without deterioration (>= 2 mm increase) of proptosis in the fellow eye.
* Proptosis relapsers: Participants who were "proptosis responders" as defined above, and then relapsed based on proptosis at any time during the 52-week follow-up period with relapse defined as follows: increase in proptosis of >= 2 mm compared to Week 16 in the study eye or deterioration of proptosis (>= 2 mm increase) in the fellow eye at any time during 52-week follow-up period.

In case of worsening of the disease, participants were allowed to receive alternative treatment for TED at the discretion of the investigator and were discontinued from the study treatment.

The primary endpoint analysis was planned to be performed once all participants had reached Week 40, which included the primary efficacy endpoint (Week 16), efficacy of retreatment for initial non-responders and relapse rates during 24 weeks of follow-up.

The final analysis was planned to be performed when the last participant had reached the end of trial.

The Food and Drug Administration (FDA) and the European Medicines Agency (EMA) expressed different preferences regarding the primary and secondary objectives and endpoints and their ordering. Therefore, this study intended to have 2 different analysis strategies and corresponding primary, secondary objective and endpoint definitions; Plan A was intended for submission in Europe (EU) and other applicable countries and Plan B was intended for submission in the United States (US) and other applicable countries. As the study was early terminated, only Plan A analysis was conducted.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient had to be able to understand and communicate with the investigator and comply with the requirements of the study and had to give a written, signed and dated informed consent before any study assessment was performed.
* Male or non-pregnant, non-lactating female patients ≥ 18 years of age.
* Clinical diagnosis of active, moderate to severe TED (not sight-threatening) in the study eye at Baseline associated with 2 or more of the following:

  * Lid retraction >= 2 mm
  * Moderate or severe soft tissue involvement
  * Exophthalmos >= 3 mm above normal
  * Inconstant or constant diplopia
* Onset of TED symptoms fewer than 12 months prior to Baseline.
* CAS >= 4 (on a 7-point scale, with a score of >= 3 indicating active TED) in the more severely affected (study) eye at Screening and Baseline. Note: Proptosis is the primary qualifier for selection of the study eye. In case both eyes showed a similar degree of proptosis, other inflammatory signs and symptoms (CAS) were taken into account by the investigator for the selection of the study eye.
* Peripheral euthyroidism or mild hypo-/hyperthyroidism defined as free T3 (fT3) and free T4 (fT4) < 30% above/below normal limits at Screening. Every effort was to be made to correct the mild hypo-/hyperthyroidism promptly and to maintain the euthyroid state until the end of this study.
* Orbital MRI assessment available confirming the diagnosis of TED for patients initially presenting with hypo- or euthyroidism (without treatment for hyperthyroidism) before or at the time of TED diagnosis (to rule out other potential causes of orbital signs and symptoms.

Key Exclusion Criteria:

* Improvement in CAS of >= 2 points and/or improvement in proptosis of >= 2 mm in the study eye between Screening and Baseline.
* Signs of sight-threatening TED defined by optic neuropathy or severe corneal injury.
* Patients, in the opinion of the investigator, requiring immediate or urgent medical treatment with glucocorticoids for TED.
* Patients requiring immediate surgical ophthalmological intervention or planning corrective surgery/irradiation during the course of the study.
* Decreased best corrected visual acuity (BCVA) as defined by a decrease in vision of 2 lines on the Snellen chart, new visual field defect or color defect within the last 6 months.
* Any other ophthalmic and/or orbital disease or condition that might interfere with the assessment of TED.
* Previous orbital radiotherapy.
* Previous ophthalmological/orbital surgery for TED (e.g., orbital decompression).
* Previous use of biological agents for the treatment of TED.
* Previous use of systemic, non-biologic, immunomodulatory agents for the treatment of TED (e.g., mycophenolate or cyclosporine).
* Previous exposure to secukinumab or other biologic drugs directly targeting IL-17A or the IL 17 receptor (e.g., ixekizumab, brodalumab).
* Previous treatment with rituximab, tocilizumab or teprotumumab.
* Previous use of systemic corticosteroids for the treatment of TED, except for oral corticosteroids with a cumulative dose equivalent to < 1 g oral prednisone/prednisolone if the corticosteroid was discontinued at least 4 weeks prior to Baseline.
* Previous treatment with any cell-depleting therapies including but not limited to anti-cluster of differentiation 20 (CD20) or investigational agents (e.g., CAMPATH, anti CD4, anti-CD5, anti-CD3, anti-CD19).
* Use of other investigational drugs within 5 half-lives of enrollment or within 30 days, whichever is longer.
* Previous or ongoing use of prohibited treatments (see Appendix 16.1.1-Protocol Section 6.2.2). Respective washout periods detailed in this section needed to be adhered to.
* History of hypersensitivity to any of the study drug constituents.

Other protocol defined Inclusion/Exclusion may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Germany (5):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Mainz

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 centers in Germany.
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio to one of the following double-blinded treatment arms: Secukinumab 300 mg (arm 1) and Placebo (arm 2).
Period: Treatment Period (Baseline to Week 16)
Arm/Group | Secukinumab 300 mg | Placebo
Started (All randomized participants were included in Full Analysis Set (FAS) and Safety Analysis Set (SAF)) | 14 | 14
Completed | 12 | 12
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Study terminated by sponsor | 1 | 2
Period: Follow-up Period (Week 16 to Week 108)
Arm/Group | Secukinumab 300 mg | Placebo
Started | 12 | 12
Completed | 8 | 9
Not Completed | 4 | 3
Not completed — Not satisfied | 1 | 0
Not completed — Study terminated by sponsor | 3 | 1
Not completed — No benefit IMP | 0 | 1
Not completed — Therapy national guidelines | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 300 mg | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (11.85) | 57.7 (10.64) | 55.6 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 5 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 14 | 28
Smoking History [Count of Participants; unit: Participants]
  Current | 3 | 4 | 7
  Former | 8 | 6 | 14
  Never | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Plan A - Percentage of Participants Achieving Overall Response
Description: The percentage of participants achieving overall response was defined as follows: >= 2 points reduction in clinical activity score (CAS) AND >= 2 mm reduction in proptosis from Baseline in the study eye, provided there was no corresponding deterioration in CAS or proptosis (>= 2 point or 2 mm increase, respectively) in the fellow eye after 16 weeks of treatment. Due to premature study discontinuation, purely descriptive analyses were performed for the primary endpoint.
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 14 | 14
Participants
  Yes | 0 | 0
  No | 12 | 11
  Missing | 2 | 3

2. Primary Outcome: Plan B - Percentage of Participants Achieving Response in Reduction of Proptosis
Description: The percentage of participants achieving response in reduction of proptosis at Week 16 was defined as follows: reduction of >= 2 mm from Baseline in the study eye without deterioration (>= 2 mm increase) of proptosis in the fellow eye. Due to premature study discontinuation, only Plan A was conducted (Plan B was not initiated) for the primary endpoint.
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS). Due to premature study discontinuation, only Plan A was conducted (no data collected for Plan B, as Plan B was not initiated).
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Plan A - Percentage of Participants Achieving Response in Reduction of Clinical Activity Score (CAS)
Description: The percentage of participants achieving response in reduction of clinical activity score (CAS) at Week 16 was defined as follows: reduction of >= 2 points from Baseline in the study eye without deterioration (>= 2 points increase) of CAS in the fellow eye. Due to premature study discontinuation, purely descriptive analyses were performed for the secondary endpoint.
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 14 | 14
Participants
  Yes | 0 | 3
  No | 12 | 8
  Missing | 2 | 3

4. Secondary Outcome: Plan A - Percentage of Participants Achieving Response in Reduction of Proptosis
Description: The percentage of participants achieving response in reduction of proptosis at Week 16 was defined as follows: reduction of >= 2 mm from Baseline in the study eye without deterioration (>= 2 mm increase) of proptosis in the fellow eye. Due to premature study discontinuation, purely descriptive analyses were performed for the secondary endpoint.
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 14 | 14
Participants
  Yes | 0 | 0
  No | 12 | 11
  Missing | 2 | 3

5. Secondary Outcome: Plan A - Percentage of Participants Achieving Response in Diplopia
Description: The percentage of participants achieving response in diplopia at Week 16 was defined as follows: Baseline diplopia > 0 and a reduction of >= 1 grade with no corresponding deterioration (>= 1 grade worsening) in the fellow eye at Week 16. Due to premature study discontinuation, purely descriptive analyses were performed for the secondary endpoint.
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 14 | 14
Participants
  Yes | 1 | 1
  No | 11 | 11
  Missing | 2 | 2

6. Secondary Outcome: Plan A - Mean Change From Baseline to Week 16 in Clinical Activity Score (CAS) in the Study Eye
Description: Thyroid Eye Disease (TED) activity was assessed using the CAS at the frequency indicated in the study schedule based on the following signs and symptoms in accordance with the European Group on Graves' Orbitopathy (EUGOGO) guideline:
  * Symptoms
    * Spontaneous retrobulbar pain
    * Pain on attempted upward or downward gaze
  * Signs
    * Redness of eyelids
    * Redness of conjunctiva
    * Swelling of caruncle or plica
    * Swelling of eyelids
    * Swelling of conjunctiva (chemosis)
  For each item present, 1 point is given. The sum of these points is the CAS score, i.e., minimum score of 0 and maximum score of 7.
  * Inactive TED: CAS < 3.
  * Active TED: CAS >= 3.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Set (FAS). Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 14 | 14
Unit on a scale
  Change from BL at Week 2 | -0.21 (0.58) | -0.29 (0.47)
  Change from BL at Week 4 | -0.14 (1.10) | -0.29 (0.73)
  Change from BL at Week 8: number analyzed (Participants) | 13 | 14
  Change from BL at Week 8 | 0.00 (1.00) | -0.21 (0.58)
  Change from BL at Week 12: number analyzed (Participants) | 12 | 14
  Change from BL at Week 12 | -0.67 (1.15) | -0.57 (0.94)
  Change from BL at Week 16: number analyzed (Participants) | 12 | 11
  Change from BL at Week 16 | 0.00 (0.95) | -0.73 (1.10)

7. Secondary Outcome: Plan A - Mean Change From Baseline to Week 16 in Millimeters (mm) of Proptosis in the Study Eye
Description: Proptosis measurements were performed at the frequency indicated in the study schedule. The same Hertel instrument, and the same outer intercanthal distance, were to be used for each measurement. The mean of measurements (change from baseline in millimeters (mm) of proptosis, calculated as: (Post-Baseline value - Baseline value) / Baseline value * 100)) for each group were presented. Due to premature study discontinuation, purely descriptive analyses were performed for the secondary endpoint.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Set (FAS). Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 14 | 14
millimeters (mm)
  Change from BL at Week 2 | 0.18 (0.72) | -0.07 (0.73)
  Change from BL at Week 4 | 0.18 (0.72) | 0.00 (1.18)
  Change from BL at Week 8: number analyzed (Participants) | 13 | 14
  Change from BL at Week 8 | 0.42 (1.00) | 0.43 (1.28)
  Change from BL at Week 12: number analyzed (Participants) | 12 | 14
  Change from BL at Week 12 | 0.67 (0.98) | 0.29 (1.33)
  Change from BL at Week 16: number analyzed (Participants) | 11 | 11
  Change from BL at Week 16 | 0.83 (1.03) | 0.64 (1.03)

8. Secondary Outcome: Plan A - Percentage of Participants With Improvement in EUGOGO Disease Severity
Description: Thyroid Eye Disease (TED) activity was assessed using the CAS at the frequency indicated in the study schedule based on the following signs and symptoms in accordance with the European Group on Graves' Orbitopathy (EUGOGO) guideline. Improvement in EUGOGO disease severity was categorized: Mild, Moderate to severe and Sight threatening.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Set (FAS). Only participants with a value at both Baseline and post-baseline visit included.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 14 | 14
Participants
  Baseline: Mild | 0 | 0
  Baseline: Moderate to severe | 14 | 14
  Baseline: Sight threatening | 0 | 0
  Week 2: Mild | 0 | 0
  Week 2: Moderate to severe | 14 | 14
  Week 2: Sight threatening | 0 | 0
  Week 4: number analyzed (Participants) | 14 | 13
  Week 4: Mild | 1 | 1
  Week 4: Moderate to severe | 13 | 12
  Week 4: Sight threatening | 0 | 0
  Week 8: number analyzed (Participants) | 13 | 14
  Week 8: Mild | 0 | 1
  Week 8: Moderate to severe | 13 | 13
  Week 8: Sight threatening | 0 | 0
  Week 12: number analyzed (Participants) | 12 | 14
  Week 12: Mild | 1 | 1
  Week 12: Moderate to severe | 11 | 13
  Week 12: Sight threatening | 0 | 0
  Week 16: number analyzed (Participants) | 12 | 11
  Week 16: Mild | 1 | 1
  Week 16: Moderate to severe | 11 | 10
  Week 16: Sight threatening | 0 | 0

9. Secondary Outcome: Plan A - Graves' Ophthalmopathy Quality of Life Questionnaire (GO-QOL) Score (Score 1: Visual Functioning) Over Time
Description: The Graves' ophthalmopathy quality of life questionnaire (GO-QOL) contains 8 questions on visual functioning and 8 questions on appearance; answers on each subscale are transformed to scores ranging from 0 (worst) to 100 (best). Due to premature study discontinuation, purely descriptive analyses were performed for the secondary endpoint.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Set (FAS). Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 14 | 14
Unit on a scale
  Baseline | 64.1 (23.04) | 66.6 (24.38)
  Week 2 | 62.9 (27.71) | 66.4 (20.51)
  Week 4 | 56.7 (28.11) | 66.7 (23.82)
  Week 8: number analyzed (Participants) | 13 | 14
  Week 8 | 51.0 (27.93) | 59.1 (24.75)
  Week 12: number analyzed (Participants) | 12 | 14
  Week 12 | 54.7 (29.45) | 60.8 (28.71)
  Week 16: number analyzed (Participants) | 12 | 11
  Week 16 | 52.1 (29.36) | 61.9 (30.42)

10. Secondary Outcome: Plan A - Graves' Ophthalmopathy Quality of Life Questionnaire (GO-QOL) Score (Score 2: Psychosocial Functioning) Over Time
Description: as for outcome 9
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Set (FAS). Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 14 | 14
Unit on a scale
  Baseline | 65.6 (22.43) | 60.3 (20.60)
  Week 2 | 68.3 (16.16) | 62.5 (29.42)
  Week 4 | 69.2 (21.01) | 56.7 (30.37)
  Week 8: number analyzed (Participants) | 13 | 14
  Week 8 | 65.4 (20.51) | 52.2 (30.87)
  Week 12: number analyzed (Participants) | 12 | 14
  Week 12 | 63.5 (26.09) | 53.1 (34.47)
  Week 16: number analyzed (Participants) | 12 | 11
  Week 16 | 66.2 (26.84) | 56.8 (30.55)

11. Secondary Outcome: Plan A - Number of Participants With Adverse Events
Description: The distribution of adverse events during Plan A study treatment period was done via the analysis of frequencies for Adverse Event (AEs) and Serious Adverse Event (SAEs), through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: From first dose of study treatment until Week 16
Population: Safety Analysis Set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 14 | 14
Participants
  Any adverse event (AE) | 9 | 6
  Study treatment related AE | 3 | 1
  AE leading to study treatment discontinuation | 0 | 0
  Serious adverse event (SAE) | 0 | 1
  Study treatment related SAE | 0 | 0
  SAE leading to study treatment discontinuation | 0 | 0

12. Secondary Outcome: Plan B - Percentage of Participants Achieving Response in Reduction of Clinical Activity Score (CAS)
Description: The percentage of participants achieving response in reduction of CAS at Week 16 was defined as follows: reduction of >= 2 points from Baseline in the study eye without deterioration (>= 2 points increase) of CAS in the fellow eye. Due to premature study discontinuation, only Plan A was conducted (Plan B was not initiated) for the secondary endpoint.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Plan B - Percentage of Participants Achieving Overall Response
Description: The percentage of participants achieving overall response was defined as follows: >= 2 points reduction in CAS AND >= 2 mm reduction in proptosis from Baseline in the study eye, provided there was no corresponding deterioration in CAS or proptosis (>= 2 point or 2 mm increase, respectively) in the fellow eye after 16 weeks of treatment. Due to premature study discontinuation, only Plan A was conducted (Plan B was not initiated) for the secondary endpoint.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Plan B - Percentage of Participants Achieving Response in Diplopia
Description: The percentage of participants achieving response in diplopia at Week 16 was defined as follows: Baseline diplopia > 0 and a reduction of >= 1 grade with no corresponding deterioration (>= 1 grade worsening) in the fellow eye at Week 16. Due to premature study discontinuation, only Plan A was conducted (Plan B was not initiated) for the secondary endpoint.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Plan B - Mean Change From Baseline to Week 16 in Clinical Activity Score (CAS) in the Study Eye.
Description: Due to premature study discontinuation, only Plan A was conducted (Plan B was not initiated) for the secondary endpoint.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Plan B - Mean Change From Baseline to Week 16 in Proptosis in the Study Eye.
Description: Proptosis is the protrusion of the eyeball. Exophthalmos means the same, and this term is usually used when describing proptosis due to Grave's disease. Due to premature study discontinuation, only Plan A was conducted (Plan B was not initiated) for the secondary endpoint.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Plan B - Mean Change From Baseline to Week 16 in the Graves' Ophthalmopathy Quality of Life Questionnaire (GO-QOL) Score (Score 1: Visual Functioning)
Description: The Graves' ophthalmopathy quality of life questionnaire (GO-QOL) contains 8 questions on visual functioning and 8 questions on appearance; answers on each subscale are transformed to scores ranging from 0 (worst) to 100 (best). Due to premature study discontinuation, only Plan A was conducted (Plan B was not initiated) for the secondary endpoint.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
Population: as for outcome 2
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Plan B - Mean Change From Baseline to Week 16 in the Graves' Ophthalmopathy Quality of Life Questionnaire (GO-QOL) Score (Score 2: Psychosocial Functioning)
Description: as for outcome 17
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
Population: as for outcome 2
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Plan B - Number of Participants With Adverse Events
Description: Due to premature study discontinuation, only Plan A was conducted (Plan B was not initiated) for the secondary endpoint.
Time Frame: From first dose of study treatment until Week 16
Population: Safety Analysis Set (SAF). Due to premature study discontinuation, only Plan A was conducted (no data collected for Plan B, as Plan B was not initiated).
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are presented for the double-blind treatment period (from first dose of study treatment until Week 16) and for the follow-up/open-label re-treatment period, including AEs in follow up for all patients who received at least one dose of Secukinumab during the entire study up to a maximum of 108 weeks.
Description: The safety analysis were done on the safety population, which included all randomized subjects who received at least one dose of study medication.
Groups:
- Secukinumab 300 mg (Double-blind): Secukinumab 300 mg (Double-blind): Double-blind treatment period (from first dose of study treatment until Week 16)
- Placebo (Double-blind): Secukinumab matching placebo (Double-blind): Double-blind treatment period (from first dose of study treatment until Week 16)
- Any Secukinumab 300 mg (Entire Study): All events reported from the beginning of the study up until the end of follow-up/open-label retreatment period (from first dose of study treatment up to Week 108)
Arm/Group | Secukinumab 300 mg (Double-blind) | Placebo (Double-blind) | Any Secukinumab 300 mg (Entire Study)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/14 | 1/26
Other Adverse Events (participants affected / at risk) | 12/14 | 12/14 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (Double-blind) (N=14) | Placebo (Double-blind) (N=14) | Any Secukinumab 300 mg (Entire Study) (N=26)
Graves' disease (Endocrine disorders) | 1 | 0 | 1
Endocrine ophthalmopathy (Eye disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (Double-blind) (N=14) | Placebo (Double-blind) (N=14) | Any Secukinumab 300 mg (Entire Study) (N=26)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Thyroid dermatopathy (Endocrine disorders) | 0 | 1 | 1
Chalazion (Eye disorders) | 0 | 1 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 0
Conjunctival oedema (Eye disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 1 | 1 | 1
Erythema of eyelid (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0
Metamorphopsia (Eye disorders) | 1 | 0 | 1
Ocular discomfort (Eye disorders) | 1 | 0 | 1
Pupillary reflex impaired (Eye disorders) | 0 | 1 | 0
Swelling of eyelid (Eye disorders) | 1 | 1 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0
Visual field defect (Eye disorders) | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 2 | 0 | 2
Injection site erythema (General disorders) | 1 | 0 | 1
Injection site haematoma (General disorders) | 0 | 1 | 1
Injection site pain (General disorders) | 1 | 0 | 1
Injection site pruritus (General disorders) | 1 | 0 | 1
Injection site swelling (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 1 | 1 | 1
Swelling (General disorders) | 0 | 1 | 0
Borrelia infection (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 4 | 6 | 10
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 0
Thyroxine free decreased (Investigations) | 1 | 0 | 1
Tri-iodothyronine increased (Investigations) | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 5
Horner's syndrome (Nervous system disorders) | 1 | 0 | 1
Acute stress disorder (Psychiatric disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT04737330/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT04737330/SAP_001.pdf